CLINICAL TRIAL: NCT01432054
Title: Human Tissue Repository for Wound Care
Status: Withdrawn | Type: Observational
Why Stopped: business decision
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: VACP2007-24
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Human Tissue Repository
Keywords: Human Tissue Repository

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — wound biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to create a Human Tissue Repository to be used as a resource for future tissue repair research at KCI USA, Inc.

DETAILED DESCRIPTION:
The study design is a multicenter study involving the collection of human biological specimens in Subjects with various wound classifications and types for the purpose of a Human Tissue Repository to be used as a resource for future tissue repair research at KCI USA, Inc. Subjects participating in this study will have a 6mm tissue punch biopsy or equivalent tissue specimen harvested from the healthiest margin of the wound. Tissue collection may occur at Visits 2, 3, 4 and 5. Visit 2 may be combined with Screening, Visit 1. Subjects will have a minimum of one (1) and a maximum of four (4) specimen collection visits. Specimens may be collected from one or multiple different tissues (connective tissue, muscle, bone, and dermis) at any or all visits. Each specimen will be placed in a separate appropriate vial. Necrotic tissue with eschar and bodily fluids such as blood, wound fluid or sputum will not be collected. Tissue from healthy, healing wounds will also be accepted. Tissue collection visits shall occur at least twenty-four (24) hours apart. Ten (10) to twenty-five (25) percent of the sites will be selected to collect all the specimens in cryovials containing a pre-aliquoted amount (1.5mL) of RNAlater. Ten (10) to twenty-five (25) percent of the sites will be selected to collect all the specimens in cryovials containing a pre-aliquoted amount of HypoThermosol. The remaining sites will collect all the specimens in a vial containing no diluents. All samples will be coded by the collection site prior to shipment to KCI.

ELIGIBILITY:
Inclusion Criteria:

* Subject's wound is acute or chronic and classified as one of the following wound types: diabetic, pressure ulcer, burn, traumatic or dehisced, and Subject signs the separate informed consent form for the study. The consent process for tissue collection should occur separately from any surgical consent.
* Subject is reported to be physically and mentally able and willing to comply with the Protocol.
* Subject is between 18 - 75 years old.

Exclusion Criteria:

* Reported presence of Human Immunodeficiency Virus.
* Reported presence of Acquired Immune Deficiency Syndrome.
* Reported presence of Hepatitis.
* Reported presence of cancer in the wound.
* Reported presence or suspected presence of infection (indicated by signs and symptoms of infection such as redness/swelling, or a positive culture, etc.)
* Presence of untreatable osteomyelitis.
* Presence of any other severe concurrent disease, which, in the judgment of the investigator, would make the subject inappropriate for entry into the study.
* Necrotic tissue with eschar present that cannot be debrided.
* Subject is unwilling or unable to comply with the protocol.
* Subject is a suspected or known intravenous drug user.
* Donation of tissue which, in the judgment of the investigator, may pose venous or arterial compromise.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects with acute or chronic wounds and whose wounds encompass one of the following wound types will be enrolled: traumatic, diabetic, pressure ulcer, burns, or dehisced wounds. Enrollment will continue up to 5 years. KCI may determine at any time that sufficient samples have been obtained and cease enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
The study design is a collection of human biological specimens in Subjects with various wound classifications and types for the purpose of a Human Tissue Repository to be used as a resource for future tissue repair research at KCI USA, Inc